CLINICAL TRIAL: NCT02134353
Title: Long Term Administration of Inhaled Mannitol in Cystic Fibrosis - A Safety and Efficacy Trial in Adult Cystic Fibrosis Subjects
Brief Title: A Safety and Efficacy Trial of Inhaled Mannitol in Adult Cystic Fibrosis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPM-CF-303
Record Dates: First submitted 2014-04-16; First posted 2014-05-09 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm A (Experimental): Active treatment. Inhaled Mannitol
  Interventions: Drug: Inhaled mannitol
- Arm B - Control (Placebo Comparator): Arm B
  Interventions: Drug: Placebo Comparator: Arm B - Control

INTERVENTIONS:
Drug: Inhaled mannitol — Inhaled mannitol 400 mg BD for 26 weeks
  Arms: Experimental arm A
Drug: Placebo Comparator: Arm B - Control — Placebo Comparator: Arm B - Control BD for 26 weeks
  Arms: Arm B - Control

SUMMARY:
This trial aims to provide prospective evidence of the safety and efficacy of mannitol 400 mg b.i.d. in subjects aged 18 years and above.

We hypothesize that inhaled mannitol 400 mg b.i.d. will increase the mean change from baseline FEV1 (mL) compared to control over the 26-week treatment period in adult subjects with cystic fibrosis. Any improvement in FEV1 is considered clinically meaningful, however, this trial has set a threshold of 80 mL for the purposes of determining an appropriate sample size for statistical power while retaining trial feasibility in an orphan disease population

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel arm, controlled, multicenter, and interventional clinical trial. Potential subjects will sign the informed consent form (ICF) and be assessed for eligibility. After satisfying all inclusion & exclusion criteria, subjects will be given a mannitol tolerance test (MTT). Those subjects that pass the MTT will be randomized to receive inhaled mannitol (400 mg b.i.d.) or control b.i.d. for a period of 26-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent to participate in this trial in accordance with local regulations;
2. Have a confirmed diagnosis of cystic fibrosis (positive sweat chloride value ≥ 60 mEq/L) and/or genotype with two identifiable mutations consistent with CF, accompanied by one or more clinical features consistent with the CF phenotype);
3. Be aged at least 18 years old;
4. Have FEV1 > 40 % and < 90% predicted (using NHanes III [1]);
5. Be able to perform all the techniques necessary to measure lung function;
6. Be adherent with maintenance therapies (antibiotics and or rhDNase), if used, for at least 80% of the time in the two weeks prior to visit 1 and
7. If rhDNase and/or maintenance antibiotic are being used treatment must have been established at least 1 month prior to screening (Visit 0). The subject should remain on the rhDNase and / or maintenance antibiotics for the duration of the trial. The subject should not commence treatment with rhDNase or maintenance antibiotics during the trial

Exclusion Criteria:

1. Be investigators, site personnel directly affiliated with this trial, or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biologically or legally adopted;
2. Be considered "terminally ill" or eligible for lung transplantation;
3. Have had a lung transplant;
4. Be using maintenance nebulized hypertonic saline in the 2 weeks prior to visit 1;
5. Have had a significant episode of hemoptysis (> 60 mL) in the three months prior to Visit 0;
6. Have had a myocardial infarction in the three months prior to Visit 0;
7. Have had a cerebral vascular accident in the three months prior to Visit 0;
8. Have had major ocular surgery in the three months prior to Visit 0;
9. Have had major abdominal, chest or brain surgery in the three months prior to Visit 0;
10. Have a known cerebral, aortic or abdominal aneurysm;
11. Be breast feeding or pregnant, or plan to become pregnant while in the trial;
12. Be using an unreliable form of contraception (female subjects at risk of pregnancy only);
13. Be participating in another investigative drug trial, parallel to, or within 4 weeks of screening (Visit 0);
14. Have a known allergy to mannitol;
15. Be using non-selective oral beta blockers;
16. Have uncontrolled hypertension -i.e. systolic BP > 190 and / or diastolic BP > 100;
17. Have a condition or be in a situation which in the Investigator's opinion may put the subject at significant risk, may confound results or may interfere significantly with the subject's participation in the trial;or
18. Have a failed or incomplete MTT at trial entry (as evaluated in Section 8.1.1.1).
19. The subject must not commence treatment with rhDNase or maintenance antibiotics during the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moira Aitken, MD, Principal Investigator; Brett Charlton, MD, Study Director — Medical Director
Locations (100):
- United States (36):
  - Dr Lawrence Sinde, Mobile, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Pediatric Pulmonology, Long Beach, California
  - University of CA, Davis, Sacramento, California
  - Hartford Hospital, Hartford, Connecticut
  - Dr Mitchell Rothstein, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cystic Fibrosis Center of Chicago, Glenview, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois Lung Institute, Peoria, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health Offices of Research Administration, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Dr Joseph Ojile, St Louis, Missouri
  - Dartmouth-Hitchcock Specialty Care, Bedford, New Hampshire
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - The Cystic Fibrosis Center Beth Israel Medical Center, New York, New York
  - Dr Allen Dozor, Valhalla, New York
  - Akron Children's Hospital, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - The Toledo Hospital and Toledo Childrens Hospital, Toledo, Ohio
  - Pediatric Pulmonary & CF Center, Oklahoma City, Oklahoma
  - Dr Santiago Reyes, Oklahoma City, Oklahoma
  - Pediatric Clinic, Portland, Oregon
  - Medical University of SC, Charleston, South Carolina
  - One Richland Medical Park, Columbia, South Carolina
  - University of Washington, Seattle, Washington
- Argentina (5):
  - Insares, Mendoza, Mendoza Province
  - Hospital Interzonal General de Agudos Dr. Jose Penna, Bahía Blanca
  - Hospital del Tórax Cetrángolo, Buenos Aires
  - Hospital Regional Español de Bahía Blanca, Buenos Aires
  - Hospital San Roque, Córdoba
- Mater Adult Hospital, Brisbane, Queensland, Australia
- Belgium (3):
  - UZ VUB, Brussels
  - UZ Leuven, Leuven
  - CHR Citadelle, Liège
- Canada (3):
  - QEII Health Sciences Center, Halifax
  - Institut de recherches cliniques de Montréal, Montreal
  - The Ottawa Hospital, General Campus, Ottawa
- FN Brno, Brno, Czechia
- Hungary (4):
  - Országos Korányi Tbc, Budapest
  - Klinikai Farmakológiai Központ, Debrecen
  - Mosdós Tüdőgyógyintézet, Mosdós
  - Törökbálint Tüdőgyógyintézet, Törökbálint
- Israel (2):
  - Pediatrics Pulmonary Department Rambam Healthcare Campus, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (7):
  - Spedali Civili Brescia, Brescia
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico Mil, Milan
  - AOU San Luigi Gonzaga, Orbassano
  - Aziendao Spedaliera Universitaria, Parma
  - Cystic Fibrosis Center Hospital San Carlo, Potenza
  - Centro Fibrosi Cistica Policlinico Umberto I, Roma
  - Azienda Ospedaliera Universitaria Integratadi Verona, Verona
- Mexico (4):
  - Instituto Jaliscience de Investigacion Clinica, Guadalajara
  - Unidad Médica de Occidente, Guadalajara
  - Arke Estudios Clinicos S.A, Mexico City
  - CEPREP- Hospital Universitario, Monterrey
- New Zealand (3):
  - Greenlane Hospital, Auckland
  - Canterbury Respiratory Research Group, Christchurch
  - Otago Respiratory Research Unit, Dunedin Hospital, Dunedin
- Poland (7):
  - Szpital Dziecięcy Polanki im. M. Płażyńskiego w Gdańsku sp., Gdansk
  - Centrum Medyczne Karpacz SA, Karpacz
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im. W. Buszkowskiego, Kielce
  - Wojewodzki Szpital Specjalistyczny im., Lodz
  - Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Sanatorium Cassia-Villa Medica S.C., Rabka-Zdrój
  - Podkarpacki Osrodek Pulmonologii i Alergologii, Rzeszów
- Romania (4):
  - Institutul pentru Ocrotirea Mamei si Copilului "Alfred Rusescu", Bucharest
  - Institutul de Pneumoftiziologie "Marius Nasta" Bucuresti, Sectia Clinica Pneumologie V, Bucharest
  - Spitalul Clinic de Pneumoftiziologie "Leon Daniello" Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie Lasi, Lasi
- Russia (5):
  - Tatiana I. Martynenko, Barnaul
  - Pulmonology Research Institute, Moscow
  - Research and Clinical Center of interstitial and orphan lung diseases, Saint Petersburg
  - Mikhail Smirnov, Vladimir
  - Clinical Hospital# 2, Yaroslavl
- Slovakia (3):
  - Oddelenie pneumológie a ftizeológie, Banská Bystrica
  - Imuno-alergologická ambulancia, Bratislava
  - Detská fakultná nemocnica Košice, Košice
- South Africa (2):
  - University of Cape Town Lung Institute, Cape Town
  - St. Augustine's Medical Centre 2, Durban
- Spain (5):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitaro La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Virgen del Rocio Hospital Unidad de Fibrosis Quistica, Seville
  - Hospital Universitario La Fe Neumología, Valencia
- Ukraine (5):
  - Dnipropetrovsk State Medical Academy, Faculty Theraphy and Endocrinology Chair, Dnipropetrovsk
  - Municipal Institution "Kherson City Clinical Hospital n.a. Afanasiy and Olha Tropin, Kherson
  - Kremenchuk First City Hospital n.a. O.T.Bogaevskyy, Kremenchuk
  - Department of Pulmonology and Thoracic Surgery of Public Institution " Kryvyy Rig City Clinical Hospital # 8, Kryvyy Rig
  - Hospital Department of Municipal Institution "Zaporizhzhya Regional Clinical Hospital", Zaporizhzhya

REFERENCES:
- [Derived] Flume PA, Amelina E, Daines CL, Charlton B, Leadbetter J, Guasconi A, Aitken ML. Efficacy and safety of inhaled dry-powder mannitol in adults with cystic fibrosis: An international, randomized controlled study. J Cyst Fibros. 2021 Nov;20(6):1003-1009. doi: 10.1016/j.jcf.2021.02.011. Epub 2021 Mar 11. PMID 33715994

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm A: Active treatment. Inhaled Mannitol
  Inhaled mannitol: Inhaled mannitol 400 mg twice a day (BD) for 26 weeks
- Arm B - Control: Arm B
  Control (mannitol 50mg) twice a day (BD) for 26 weeks
Period: Overall Study
Arm/Group | Experimental Arm A | Arm B - Control
Started | 209 | 214
Completed | 183 | 190
Not Completed | 26 | 24
Not completed — Adverse Event | 10 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Withdrawal by Subject | 12 | 13
Not completed — Death | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Relocation | 1 | 0
Not completed — Other - Patient's Choice | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT - all patients randomised
Groups:
- Arm B - Control: Arm B
  Control BD (mannitol 50mg) for 26 weeks
- Total: Total of all reporting groups
Arm/Group | Experimental Arm A | Arm B - Control | Total
Number analyzed (Participants) | 209 | 214 | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (7.63) | 28.6 (10.75) | 27.7 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 107 | 199
  Male | 117 | 107 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 7 | 21
  Not Hispanic or Latino | 195 | 207 | 402
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 202 | 209 | 411
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Argentina | 4 | 2 | 6
  Romania | 5 | 5 | 10
  Hungary | 9 | 8 | 17
  United States | 57 | 59 | 116
  Czechia | 0 | 1 | 1
  Ukraine | 31 | 32 | 63
  Russia | 21 | 20 | 41
  Spain | 6 | 5 | 11
  New Zealand | 2 | 3 | 5
  Canada | 7 | 6 | 13
  Belgium | 3 | 3 | 6
  Poland | 22 | 22 | 44
  Italy | 7 | 8 | 15
  Mexico | 3 | 2 | 5
  South Africa | 4 | 6 | 10
  Slovakia | 8 | 9 | 17
  Israel | 4 | 7 | 11
  Australia | 2 | 2 | 4
  Bulgaria | 6 | 7 | 13
  Greece | 4 | 3 | 7
  Turkey | 4 | 4 | 8
%Predicted FEV1 at Screening [Count of Participants; unit: Participants] — FEV1 (forced expiratory volume at one second)
  Participants
    >80% to <=90% | 31 | 27 | 58
    >70% to <=80% | 54 | 52 | 106
    >40% to <=70% | 124 | 135 | 259
CFTR Mutation [Count of Participants; unit: Participants] — CFTR (cystic fibrosis transmembrane conductance regulator) Mutation
  Participants
    Both deltaF508 | 55 | 48 | 103
    One deltaF508 | 91 | 89 | 180
    At least one other known mutation | 28 | 37 | 65
    Both unknown | 35 | 40 | 75
Hospitalisations due to exacerbations in 12 months prior to screening [Count of Participants; unit: Participants]
  0 | 121 | 135 | 256
  1 | 57 | 43 | 100
  2 | 20 | 23 | 43
  3 | 11 | 9 | 20
  4 | 0 | 3 | 3
  >4 | 0 | 1 | 1
Exacerbations treated with IV antibiotics in 12 months before screening [Count of Participants; unit: Participants]
  0 | 109 | 120 | 229
  1 | 58 | 47 | 105
  2 | 28 | 32 | 60
  3 | 13 | 11 | 24
  4 | 1 | 3 | 4
  >4 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in FEV1 (mL) From Baseline (Visit 1) Over the 26-week Treatment Period (to Visit 4).
Description: The mean absolute change from baseline FEV1 (mL) over 26 weeks (measured at week 6, 14 and 26) will be compared between the two treatment groups with a REML (restricted maximum likelihood) based repeated measures approach.
  Least square means presented are for the average change over the 6, 14, and 26 week visits.
  Missing values due to withdrawal for reasons related to safety or efficacy were imputed using a baseline observation carried forward approach (BOCF).
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
mL | 63 [25 to 100] | 8 [-27 to 44]
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.020, Mixed Models Analysis; Mean Difference (Net) = 54, 95% CI 2-sided [8 to 100] — Missing data for withdrawals related to safety or efficacy imputed using BOCF (baseline observation carried forward). Data collected at 6, 14 and 26 weeks

2. Secondary Outcome: Mean Change From Baseline FVC (mL) Over the 26-week Treatment Period
Description: To determine whether inhaled mannitol (400 mg b.i.d.) is superior to control for improving lung function as measured by mean change from baseline forced vital capacity (FVC) (mL) over the 26-week treatment period in adult subjects with cystic fibrosis (CF).
  The mean absolute change from baseline FVC (mL) over 26 weeks will be compared between the two treatment groups with a REML (restricted maximum likelihood) based repeated measures approach.
  Least square means presented are for the change from baseline averaged over the treatment period (ie the average of the changes at 6 weeks, 14 weeks and 26 weeks).
  Missing values due to withdrawal for reasons related to safety or efficacy were imputed using a baseline observation carried forward approach (BOCF).
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
mL | 28 [-14 to 70] | -12 [-53 to 29]
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.128, Mixed Models Analysis — Missing data for withdrawals due to safety/efficacy imputed using BOCF. Data collected at 6,14 and 26 weeks; Mean Difference (Net) = 40, 95% CI 2-sided [-12 to 92] — Missing data for withdrawals related to safety or efficacy imputed using BOCF. Data collected at 6, 14 and 26 weeks

3. Other Pre Specified Outcome: Time to First Pulmonary Exacerbation Over the 26-week Treatment Period
Description: To determine whether inhaled mannitol (400 mg b.i.d.) is superior to control in increasing the time to first protocol defined pulmonary exacerbation over the 26-week treatment period in adult subjects with CF.
  Protocol defined pulmonary exacerbations are those where 4 or more symptoms are recorded and are treated with IV antibiotics
Time Frame: 26 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
days | NA [NA to NA] — Too few participants with protocol defined pulmonary exacerbations (PDPE), median time to first PDPE not reached | NA [NA to NA] — Too few participants with protocol defined pulmonary exacerbations (PDPE), median time to first PDPE not reached
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.629, Regression, Cox; Cox Proportional Hazard = 1.140, 95% CI 2-sided [0.671 to 1.936]

4. Other Pre Specified Outcome: Number of Days on Antibiotics (Oral, Inhaled or IV) Due to Pulmonary Exacerbation
Description: To determine whether in adult subjects with CF, inhaled mannitol (400 mg b.i.d.) is superior to control for decreasing the number of days on antibiotics due to protocol defined pulmonary exacerbations.
  Overlapping antibiotics are counted separately.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
days | 8.1 (31.25) | 5.5 (17.94)
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.673, Negative binomial model; Rate ratio = 0.750, 95% CI 2-sided [0.198 to 2.846]

5. Other Pre Specified Outcome: Number of Days in Hospital Due to Pulmonary Exacerbation
Description: To determine whether in adult subjects with CF, inhaled mannitol (400 mg b.i.d.) is superior to control for decreasing the number of days in hospital due to protocol defined pulmonary exacerbation.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
Participants
  0 days | 192 | 199
  1-7 days | 1 | 4
  8-14 days | 4 | 6
  15-21 days | 5 | 3
  22-28 days | 3 | 2
  >28 days | 4 | 0
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.735, Negative binomial model; Rate ratio = 1.273, 95% CI 2-sided [0.315 to 5.154]

6. Other Pre Specified Outcome: Rate of Pulmonary Exacerbations Over the 26-week Treatment Period
Description: To determine whether inhaled mannitol (400 mg b.i.d.) decreases the rate of protocol defined pulmonary exacerbations over the 26-week treatment period compared to control in adult subjects with CF.
  Protocol defined pulmonary exacerbations defined by having 4 or more symptoms and treated with IV antibiotics.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
Participants
  0 protocol defined pulm exac | 181 | 185
  1 protocol defined pulm exac | 24 | 29
  2 protocol defined pulm exac | 3 | 0
  >2 protocol defined pulm exac | 1 | 0
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Patients withdrawing early without an exacerbation had rate imputed based on number of exacerbations in 12 months prior to screening; Test type: Superiority; p = 0.055, Negative binomial model; Rate ratio = 1.545, 95% CI 2-sided [0.990 to 2.411]
Statistical Analysis 2: Comparison: Experimental Arm A vs Arm B - Control; Sensitivity analysis with no imputation of missing data; Test type: Superiority; p = 0.246, Negative binomial model; Rate ratio = 1.357, 95% CI 2-sided [0.810 to 2.275]

7. Other Pre Specified Outcome: The Incidence of Pulmonary Exacerbations
Description: To determine whether in adult subjects with CF, inhaled mannitol (400 mg b.i.d.) is superior to control for decreasing incidence of protocol defined pulmonary exacerbations, where incidence is defined as the proportion of subjects with 1 or more exacerbation during the 26 week period.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
Participants | 28 | 29
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.976, Regression, Logistic; Odds Ratio (OR) = 1.009, 95% CI 2-sided [0.555 to 1.836]

8. Other Pre Specified Outcome: Mean Change From Baseline in Ease of Expectoration Measured Using a Visual Analogue Scale (VAS) Over 26 Weeks
Description: To determine whether in adult subjects with CF, inhaled mannitol (400 mg b.i.d.) is superior to control for improving ease of expectoration.
  The visual analogue scale (VAS) was 10cm. The position marked by the subject was converted into a score from 0 to 100 where 0 was the worst possible outcome and 100 was the best possible outcome.
  The VAS was completed at baseline, 6, 14 and 26 weeks. The mean absolute change from baseline over 26 weeks (ie the average of the changes at 6,14 and 26 weeks) is the outcome measure and will be compared between the two treatment groups with a REML based repeated measures approach.
  Least square means presented are for the change from baseline averaged over the treatment period (ie the average of the changes at 6 weeks, 14 weeks and 26 weeks).
  Missing values due to withdrawal for reasons related to safety or efficacy were imputed using a baseline observation carried forward approach (BOCF).
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
cm | 0.795 [0.556 to 1.034] | 0.537 [0.306 to 0.767]
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.083, Mixed Models Analysis; Missing values due to withdrawal related to safety/efficacy imputed using BOCF; Mean Difference (Net) = 0.259, 95% CI 2-sided [-0.034 to 0.551]

9. Other Pre Specified Outcome: Change From Baseline Over 26 Weeks in CFQ-R Respiratory Domain Score
Description: To determine whether in adult subjects with CF, inhaled mannitol (400 mg b.i.d.) is superior to control for improving respiratory symptoms measured by Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory domain.
  The CFQ-R respiratory domain score is a scale from 0 to 100. Higher scores are a more favourable response.
  The mean absolute change from baseline over 26 weeks (measured at week 6, 14 and 26) will be compared between the two treatment groups with a REML (restricted maximum likelihood) based repeated measures approach.
  Least square means presented are for the change from baseline averaged over the treatment period (ie the average of the changes at 6 weeks, 14 weeks and 26 weeks).
  Missing values due to withdrawal for reasons related to safety or efficacy were imputed using a baseline observation carried forward approach (BOCF).
Time Frame: 26 weeks
Population: Intent to Treat (ITT) - All patients randomised.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
score on a scale | 0.308 [-1.554 to 2.169] | -0.562 [-2.357 to 1.234]
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.453, Mixed Models Analysis; Mean Difference (Net) = 0.870, 95% CI 2-sided [-1.406 to 3.145] — Missing values due to withdrawal related to safety/efficacy imputed using BOCF

10. Post Hoc Outcome: Absolute Change in Forced Expiratory Flow From 25% to 75% of Vital Capacity (FEF25-75) Over the 26-week Treatment Period.
Description: The mean absolute change from baseline FEF25-75 (mL/s) over weeks 6, 14 and 26 will be compared between the two treatment groups with a REML based repeated measures approach
  Least square means presented are for the change from baseline averaged over the treatment period (ie the average of the changes at 6 weeks, 14 weeks and 26 weeks).
  Missing values due to withdrawal for reasons related to safety or efficacy were imputed using a baseline observation carried forward approach (BOCF).
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/s
Arm/Group | Experimental Arm A | Arm B - Control
Number analyzed (Participants) | 209 | 214
mL/s | 109 [54 to 164] | 22 [-32 to 75]
Statistical Analysis 1: Comparison: Experimental Arm A vs Arm B - Control; Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Net) = 87, 95% CI 2-sided [20 to 155] — Missing data due to withdrawals for reasons related to safety/efficacy imputed using BOCF

ADVERSE EVENTS:
Time Frame: 26 weeks
Groups:
- Experimental Arm A: Active treatment. Inhaled Mannitol
  Inhaled mannitol: Inhaled mannitol 400 mg BD for 26 weeks
  Subjects randomised and treated.
- Arm B - Control: Arm B
  Control BD (mannitol 50mg) for 26 weeks
  Subjects randomised and treated.
Arm/Group | Experimental Arm A | Arm B - Control
All-Cause Mortality (participants affected / at risk) | 0/207 | 1/213
Serious Adverse Events (participants affected / at risk) | 31/207 | 29/213
Other Adverse Events (participants affected / at risk) | 144/207 | 140/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm A (N=207) | Arm B - Control (N=213)
Condition Aggravated (General disorders) | 20 (25) | 15 (15) — Pulmonary exacerbations were coded to condition aggravated
Lung Infection (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm A (N=207) | Arm B - Control (N=213)
Condition Aggravated (General disorders) | 56 (84) | 59 (75) — Pulmonary Exacerbations coded as condition aggravated Includes both serious and non-serious AEs (separate summaries of non-serious AEs not available)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 21 (25)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 (27) | 20 (33)
Headache (Nervous system disorders) | 12 (41) | 22 (47)
Upper Respiratory Tract Infection (Infections and infestations) | 14 (17) | 11 (12)
Pyrexia (General disorders) | 13 (18) | 8 (9)
Nasopharyngitis (Infections and infestations) | 12 (17) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT02134353/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT02134353/SAP_001.pdf